CLINICAL TRIAL: NCT00957580
Title: Phase II Trial With Safety-Run-In of MEK Inhibitor MSC1936369B in Subjects With Poor Prognosis Acute Myeloid Leukemia and Other Hematological Malignancies
Brief Title: Trial of Pimasertib in Hematological Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial has been terminated due to an estimated low probability of clinical benefit based on limited anti-leukemic effects observed in safety run-in (Part 1)
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR200066_002; 2009-010866-49 (EudraCT Number)
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Leukemia, Myeloid, Acute; Hematologic Neoplasms
Keywords: MEK Inhibitor; Pimasertib; Acute Myeloid Leukemia; Hematological Malignancies; Elderly Patients; Phase II
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Hematologic Neoplasms | interventions — N-(2,3-dihydroxypropyl)-1-((2-fluoro-4-iodophenyl)amino)isonicotinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Regimen 1 (Part 1) (Experimental)
  Interventions: Drug: Pimasertib
- Regimen 2 (Part 1) (Experimental)
  Interventions: Drug: Pimasertib
- Regimen 3 (Part 1) (Experimental)
  Interventions: Drug: Pimasertib
- Regimen 1 (Part 2) (Experimental)
  Interventions: Drug: Pimasertib
- Regimen 2 (Part 2) (Experimental)
  Interventions: Drug: Pimasertib

INTERVENTIONS:
Drug: Pimasertib — Pimasertib will be administered orally at a dose of 8 mg twice daily (BID) on Days 1 to 5, 8 to 12, 15 to 19, and 22 to 26 of a 28-day cycle. The dose will be escalated to 15 mg BID, 23 mg BID, 30 mg BID, 42 mg BID, 60 mg BID, and 75 mg BID) until Maximum Tolerated Dose (MTD) is reached. The treatment will be continued until disease progression, intolerable toxicity, or Investigator/subject decision.
  Other Names: MSC1936369B
  Arms: Regimen 1 (Part 1)
Drug: Pimasertib — Pimasertib will be administered orally at a dose of 8 mg BID on Days 1 to 21 of a 28-day cycle. The dose will be escalated to 15 mg BID, 23 mg BID, 30 mg BID, 42 mg BID, 45 mg BID, 60 mg BID, 75 mg BID, and 90 mg BID until MTD is reached. The treatment will be continued until disease progression, intolerable toxicity, or Investigator/subject decision.
  Other Names: MSC1936369B
  Arms: Regimen 2 (Part 1)
Drug: Pimasertib — Pimasertib will be administered orally at a dose of 60 mg BID on Days 1-28 of a 28-day cycle. The dose escalation will proceed to 75 mg BID until MTD is reached. The treatment will be continued until disease progression, intolerable toxicity, or Investigator/subject decision.
  Other Names: MSC1936369B
  Arms: Regimen 3 (Part 1)
Drug: Pimasertib — Pimasertib will be administered orally twice daily on Days 1 to 5, 8 to 12, 15 to 19, and 22 to 26 of a 28-day cycle. Dose will be determined by Part 1 of the trial (could be the MTD or lower dose level). The treatment will be continued until disease progression, intolerable toxicity, or Investigator/subject decision.
  Other Names: MSC1936369B
  Arms: Regimen 1 (Part 2)
Drug: Pimasertib — Pimasertib will be administered orally twice daily on Days 1 to 21 of a 28-day cycle. Dose will be determined by Part 1 of the trial (could be the MTD or lower dose level). The treatment will be continued until disease progression, intolerable toxicity, or Investigator/subject decision.
  Other Names: MSC1936369B
  Arms: Regimen 2 (Part 2)

SUMMARY:
This is an open-label, multi-center, dose-escalation trial of pimasertib (MSC1936369B) in blood and bone marrow cancers. The trial will be conducted in two parts:

Part 1 (safety run-in period): Will determine the maximum tolerated dose (MTD) of the study drug in subjects with advanced hematological malignancies.

Part 2: Will assess the anti-leukemic activity of the study drug in older subjects with newly diagnosed poor prognosis acute myeloid leukemia (AML) who are not candidates for intensive chemotherapy.

ELIGIBILITY:
Inclusion criteria:

Part 1:

1. Subjects with one of the following conditions:

   * Primary or secondary AML, pathologically confirmed according to World Health Organization (WHO) classification who meet at least one of the following conditions:

     1. Subjects with second or subsequent relapse after standard therapy, for whom no established treatment options are available
     2. Subjects refractory to available therapies, for example, who failed to achieve complete response (CR) after 2 induction chemotherapy treatments
     3. Newly-diagnosed older subjects (greater than or equal to 75 years of age), not candidates for intensive chemotherapy
   * Subjects with myelodysplastic syndrome (MDS), International Prognostic Scoring System (IPSS) Int-2 or high risk who are resistant or intolerant to standard treatment and not candidates for transplantation
   * Subjects with relapsed or refractory multiple myeloma (MM), who have failed or are intolerant to at least two prior therapies including thalidomide, lenalidomide and bortezomib
   * Subjects with advanced myeloproliferative disorders (MPD) for whom no established treatment options are available
   * Subjects with acute lymphocytic leukemia (ALL), relapsed, refractory or intolerant to standard treatment and for whom no effective treatment options are available
2. Age greater than or equal to 18 years
3. Subjects have read and understood the Informed Consent Form and are willing and able to give informed consent. They fully understand requirements of the trial and are willing to comply with all trial visits and assessments
4. Subjects and their partners must be willing to avoid pregnancy during the trial and until 1 month after the last trial drug administration. Subjects must therefore be willing to use adequate contraception as approved by the Investigator, two barrier methods or one barrier method with spermicide or intrauterine device, 2 weeks before, during the trial and 1 month after. The use of hormonal contraceptives should be avoided due to a possible drug-drug interaction in female subjects of childbearing age

Part 2:

1. Subjects (male and female) with newly diagnosed primary or secondary AML pathologically confirmed according to WHO classification who have not been exposed to any prior therapy for AML with the exception of:

   * Emergency leukapheresis and
   * Emergency treatment for hyperleukocytosis with hydroxyurea that is allowed until 24 hours before the start of the trial treatment. Prior therapy for pre-existing hematological conditions, for example, MDS or MPD, including but not limited to hypomethylating agents, is also allowed until at least 2 weeks or 5 half-lives of that agent before the first dose of pimasertib
2. Subjects meet at least one of the following conditions:

   * Age greater than or equal to 75 years OR
   * Age greater than or equal to 60 and less than 75 years with at least one of the following poor prognostic factors:

     * Secondary AML, as determined by known and documented exposure to leukemogenic therapy or environmental toxin or antecedent history of MDS or MPD according to WHO criteria for at least 3 months prior to trial entry, with prior bone marrow aspirate, biopsy and peripheral blood smear documenting the diagnosis
     * At least one of the following unfavorable cytogenetic abnormalities: del(5q), -5, -7, del(7q), abn 3q, 9q, 11q, 20q, 21q, 17p, t(6;9), t(9;22) or complex karyotypes (greater than or equal to 3 unrelated abnormalities)
     * Eastern Cooperative Oncology Group (ECOG) status 2
3. Subjects have read and understood the Informed Consent Form and are willing and able to give informed consent. They fully understand requirements of the trial and are willing to comply with all trial visits and assessments
4. Subjects and their partners must be willing to avoid pregnancy during the trial and until 1 month after the last trial drug administration. Subjects must therefore be willing to use adequate contraception as approved by the Investigator such as two barrier methods or one barrier method with spermicide or intrauterine device, 2 weeks before, during the trial and 1 month after. The use of hormonal contraceptives should be avoided due to a possible drug-drug interaction in female subjects of childbearing age

Exclusion Criteria:

Part 1 and Part 2:

1. ECOG performance status 3 or greater
2. Hyperleukocytosis with greater than 30 x 10 to the ninth power per liter leukemia blasts in peripheral blood
3. Acute promyelocytic leukemia [t(15;17)]
4. Administration of any antineoplastic therapy within at least 2 weeks or 5 half lives of that therapy of the first pimasertib dose; except the use of hydroxyurea as permitted in inclusion criteria
5. Participation in other clinical trials within at least 2 weeks of the first pimasertib dose
6. Clinical evidence of active central nervous system leukemia
7. Active and uncontrolled infection including but not limited to known infection with human immunodeficiency virus (HIV), active hepatitis B or hepatitis C. Subjects with an infection receiving treatment with antibiotics may be entered into the trial if they are afebrile and hemodynamically stable for 48 hours prior to trial entry
8. Major surgery within two weeks prior to trial entry
9. Liver function tests above the following limits at screening: total bilirubin >1.5 x upper limit of normal (ULN) unless related to Gilbert's syndrome or hemolysis, aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >2.5 x ULN, or for subjects with liver involvement AST and/or ALT >5 x ULN
10. Serum creatinine >1.5 x ULN and /or creatinine clearance <30 milliliter per minute (mL/min) at screening
11. International normalized ratio (INR) greater than 1.5 x ULN unless on treatment with warfarin
12. For female subjects: pregnant or breast-feeding
13. History of difficulty swallowing, malabsorption or other chronic gastro-intestinal disease or conditions that may hamper compliance and/or absorption of the tested product
14. Has significant cardiac conduction abnormalities and/or pacemaker
15. Has retinal degenerative disease (heredity retinal degeneration or age-related macular degeneration), history of uveitis or history of retinal vein occlusion and/or any medically relevant abnormal findings at the initial ophthalmologic examination
16. Subjects with solid tumors, for whom the Investigator has clinical suspicion of active disease at the time of enrolment. Subjects with adequately treated early stage squamous cell carcinoma of the skin, basal cell carcinoma of the skin, or cervical intraepithelial neoplasia (CIN) are eligible for this study
17. Signs and symptoms suggestive of transmissible spongiform encephalopathy, or family members who suffer(ed) from such
18. Other significant disease that in the Investigator's opinion would exclude the subject from the trial
19. Legal incapacity or limited legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-09-30 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (9):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
- France (4):
  - Hospital Hotel Dieu, Service D'Hematologie, Nantes, Cedex
  - Hospital Edouard Herriot, Service d'Hematologie Clinique, Lyon
  - Hospital Saint Louis, Service des Maladies du Sang, Paris
  - CHU du Haut-Leveque, Service des Maladies du Sang Unite de Recherche Clinique, Pessac

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last subject (informed consent): September 2009/12 April 2012. Last subject completed : December 2012; Clinical data cut-off: December 2012.
Pre-assignment Details: Enrolled: 116 screened for eligibility; 35 were excluded (mainly non-fulfillment of inclusion or exclusion). 81 subjects were randomized.
Groups:
- Regimen 1 (Part 1): Pimasertib was administered orally at a dose of 8 mg twice daily (BID) on Days 1 to 5, 8 to 12, 15 to 19, and 22 to 26 of a 28-day cycle. The dose was escalated to 15 mg BID, 23 mg BID, 30 mg BID, 42 mg BID, 60 mg BID, and 75 mg BID) until Maximum Tolerated Dose (MTD) was obtained. The treatment was continued until disease progression, intolerable toxicity, or Investigator/subject decision.
- Regimen 2 (Part 1): Pimasertib was administered orally at a dose of 8 mg BID on Days 1 to 21 of a 28-day cycle. The dose was escalated to 15 mg BID, 23 mg BID, 30 mg BID, 42 mg BID, 45 mg BID, 60 mg BID, 75 mg BID, and 90 mg BID until MTD was obtained. The treatment was continued until disease progression, intolerable toxicity, or Investigator/subject decision.
- Regimen 3 (Part 1): Pimasertib was administered orally at a dose of 60 mg BID on Days 1-28 of a 28-day cycle. The dose was escalated to 75 mg BID until MTD was obtained. The treatment was continued until disease progression, intolerable toxicity, or Investigator/subject decision.
Period: Overall Study
Arm/Group | Regimen 1 (Part 1) | Regimen 2 (Part 1) | Regimen 3 (Part 1)
Started | 33 | 33 | 15
Treated | 33 | 32 | 15
Completed | 33 | 31 | 15
Not Completed | 0 | 2 | 0
Not completed — Ongoing at data cut-off | 0 | 1 | 0
Not completed — Enrolled but not treated | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all the subjects who were treated with at least one administration of pimasertib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen 1 (Part 1) | Regimen 2 (Part 1) | Regimen 3 (Part 1) | Total
Number analyzed (Participants) | 33 | 32 | 15 | 80
Age, Customized [Number; unit: Subjects]
  18 to less than (<) 60 | 14 | 12 | 6 | 32
  60 to <75 | 13 | 16 | 6 | 35
  Greater than or equal to (>=) 75 | 6 | 4 | 3 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 7 | 29
  Male | 24 | 19 | 8 | 51

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Subjects With Dose Limiting Toxicities (DLTs)
Description: The DLT was any toxicity that resulted in treatment delay for more than (>) 2 weeks due to treatment-related adverse effects, or any Grade greater than or equal to (>=) 3 non-hematological toxicity excluding Grade 4 asymptomatic increases in liver function tests reversible within 7 days in subjects with liver involvement, and Grade 3 asymptomatic increases in liver function tests reversible within 7 days for subjects without liver involvement, Grade 3 vomiting unless encountered and persistent for more than 3 days despite adequate and optimal therapy, and Grade 3 diarrhea unless encountered and persistent for more than 3 days despite adequate and optimal anti-diarrhea therapy at any DL and judged to be possibly or probably related to the trial treatment by the Investigator and/or the Sponsor.
Time Frame: Baseline Up to Day 29 of Cycle 1
Population: The DLT analysis set included all subjects who received over 90 percent (%) administration of trial medication in Cycle 1 or showed a DLT.
Measure: Number; unit: subjects
Arm/Group | Regimen 1 (Part 1) | Regimen 2 (Part 1) | Regimen 3 (Part 1)
Number analyzed (Participants) | 21 | 22 | 13
subjects | 1 | 0 | 5

2. Primary Outcome: Part 2: Percentage of Subjects With Best Overall Response
Description: The best overall response was to be reported as either of the following: (1) Morphologic complete remission (CR) = normalization of the peripheral blood absolute neutrophil count (PBANC) >1.0x10^9 per liter (/L), platelets >100x10^9 /L, bone marrow aspirate with less than or equal to (<=) 5 percent (%) blasts, no blasts with Auer rods (AML only). (2) Complete remission with incomplete blood count recovery (CRi) = Same as CR without normalization of PBANC and platelet count. (3) Partial remission (PR) = normalization of PBANC >1.0x10^9/L, platelets >100x10^9/L, and at least a 50% decrease in the percentage of marrow aspirate blasts to 5-25%, or marrow blasts less than (<) 5%. (4) Progressive disease (PD) = >50% increase in peripheral blood or bone marrow blasts. (5) Stable disease (SD) = subjects who failed to achieve CR, CRi or PR and without criteria for PD.
Time Frame: Day 29 of every 29-day cycle until progression reported between day of first subject randomized, September 2009, until cut-off date, December 2012
Population: Due to limited anti-leukemic effects observed in the safety run-in part decision was made not to conduct part 2 hence this outcome measure was not assessed. Effects observed in the safety run-in part decision was made not to conduct part 2 hence this outcome measure was not assessed.
Groups:
- Regimen 1 (Part 2): Pimasertib was to be administered orally twice daily on Days 1 to 5, 8 to 12, 15 to 19, and 22 to 26 of a 28-day cycle. Dose was to be determined by Part 1 of the trial (could be the MTD or lower dose level). The treatment was to be continued until disease progression, intolerable toxicity, or Investigator/subject decision.
- Regimen 2 (Part 2): Pimasertib was to be administered orally twice daily on Days 1 to 21 of a 28-day cycle. Dose was to be determined by Part 1 of the trial (could be the MTD or lower dose level). The treatment was to be continued until disease progression, intolerable toxicity, or Investigator/subject decision.
Arm/Group | Regimen 1 (Part 2) | Regimen 2 (Part 2)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Part 1: Number of Subjects With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Death and TEAEs Leading to Permanent Treatment Discontinuation
Description: An adverse event (AE) was defined as any new untoward medical occurrences/worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs include both SAEs and non-SAEs.
Time Frame: Baseline up to 3 years
Population: The safety analysis set included all the subjects who received at least one administration of the trial medication.
Measure: Number; unit: Subjects
Arm/Group | Regimen 1 (Part 1) | Regimen 2 (Part 1) | Regimen 3 (Part 1)
Number analyzed (Participants) | 33 | 32 | 15
Subjects
  TEAEs | 33 | 32 | 15
  Serious TEAEs | 24 | 28 | 12
  TEAEs Leading to Death | 6 | 6 | 5
  TEAEs Leading to Treatment Discontinuation | 7 | 7 | 7

4. Secondary Outcome: Part 1: Maximum Plasma Concentration (Cmax) of Pimasertib Single Dose
Time Frame: Predose 0.5, 1.0, 1.5, 2.0, 2.5, 4.0, 6.0, and 10.0 hours post-dose on Day 1 of cycle 1; Regimen 1, 2 and 3
Population: Pharmacokinetic analysis set included all the subjects who received at least 1 dose of trial medication and provided adequate PK samples per protocol. N (number of subject analyzed) signifies subjects evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter
Groups:
- Pimasertib 8 mg (All Regimens [Part 1]): Pimasertib was administered orally at a dose of 8 mg twice daily (BID) on Days 1 to 5, 8 to 12, 15 to 19, and 22 to 26 of a 28-day cycle in Regimen 1; and on Days 1 to 21 of a 28-day cycle in Regimen 2. The treatment was continued until disease progression, intolerable toxicity, or Investigator/subject decision.
- Pimasertib 15 mg (All Regimens [Part 1]): Pimasertib was administered orally at a dose of 15 mg twice daily (BID) on Days 1 to 5, 8 to 12, 15 to 19, and 22 to 26 of a 28-day cycle in Regimen 1; and on Days 1 to 21 of a 28-day cycle in Regimen 2. The treatment was continued until disease progression, intolerable toxicity, or Investigator/subject decision.
- Pimasertib 23 mg (All Regimens [Part 1]): Pimasertib was administered orally at a dose of 23 mg twice daily (BID) on Days 1 to 5, 8 to 12, 15 to 19, and 22 to 26 of a 28-day cycle in Regimen 1; and on Days 1 to 21 of a 28-day cycle in Regimen 2. The treatment was continued until disease progression, intolerable toxicity, or Investigator/subject decision.
- Pimasertib 30 mg (All Regimens [Part 1]): Pimasertib was administered orally at a dose of 30 mg twice daily (BID) on Days 1 to 5, 8 to 12, 15 to 19, and 22 to 26 of a 28-day cycle in Regimen 1; and on Days 1 to 21 of a 28-day cycle in Regimen 2. The treatment was continued until disease progression, intolerable toxicity, or Investigator/subject decision.
- Pimasertib 42 mg (All Regimens [Part 1]): Pimasertib was administered orally at a dose of 42 mg twice daily (BID) on Days 1 to 5, 8 to 12, 15 to 19, and 22 to 26 of a 28-day cycle in Regimen 1; and on Days 1 to 21 of a 28-day cycle in Regimen 2. The treatment was continued until disease progression, intolerable toxicity, or Investigator/subject decision.
- Pimasertib 45 mg (All Regimens [Part 1]): Pimasertib was administered orally at a dose of 45 mg twice daily (BID) on Days 1 to 21 of a 28-day cycle in Regimen 2. The treatment was continued until disease progression, intolerable toxicity, or Investigator/subject decision.
- Pimasertib 60 mg (All Regimens [Part 1]): Pimasertib was administered orally at a dose of 60 mg twice daily (BID) on Days 1 to 5, 8 to 12, 15 to 19, and 22 to 26 of a 28-day cycle in Regimen 1; on Days 1 to 21 of a 28-day cycle in Regimen 2; and on Days 1-28 of a 28-day cycle in Regimen 3. The treatment was continued until disease progression, intolerable toxicity, or Investigator/subject decision.
- Pimasertib 75 mg (All Regimens [Part 1]): Pimasertib was administered orally at a dose of 75 mg twice daily (BID) on Days 1 to 5, 8 to 12, 15 to 19, and 22 to 26 of a 28-day cycle in Regimen 1; on Days 1 to 21 of a 28-day cycle in Regimen 2; and on Days 1-28 of a 28-day cycle in Regimen 3. The treatment was continued until disease progression, intolerable toxicity, or Investigator/subject decision.
- Pimasertib 90 mg (All Regimens [Part 1]): Pimasertib was administered orally at a dose of 90 mg twice daily (BID) on Days 1 to 21 of a 28-day cycle in Regimen 2. The treatment was continued until disease progression, intolerable toxicity, or Investigator/subject decision.
Arm/Group | Pimasertib 8 mg (All Regimens [Part 1]) | Pimasertib 15 mg (All Regimens [Part 1]) | Pimasertib 23 mg (All Regimens [Part 1]) | Pimasertib 30 mg (All Regimens [Part 1]) | Pimasertib 42 mg (All Regimens [Part 1]) | Pimasertib 45 mg (All Regimens [Part 1]) | Pimasertib 60 mg (All Regimens [Part 1]) | Pimasertib 75 mg (All Regimens [Part 1]) | Pimasertib 90 mg (All Regimens [Part 1])
Number analyzed (Participants) | 9 | 6 | 9 | 7 | 9 | 4 | 19 | 10 | 4
nanogram/milliliter | 14.8 (43.0) | 29.3 (32.0) | 59.1 (86.2) | 132.8 (29.6) | 151.6 (38.8) | 207.0 (27.8) | 269.9 (46.1) | 241.9 (81.0) | 342.6 (18.5)

5. Secondary Outcome: Part 1: Maximum Plasma Concentration (Cmax) of Pimasertib Multiple Dose
Time Frame: Pre dose 0.5, 1.0, 1.5, 2.0, 2.5, 4.0, 6.0, and 10.0 hours post dose in Cycle 1 on Day 19 to Day 21 (Regimen 1 and 2) or Day 26 (Regimen 3).
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter
Arm/Group | Pimasertib 8 mg (All Regimens [Part 1]) | Pimasertib 15 mg (All Regimens [Part 1]) | Pimasertib 23 mg (All Regimens [Part 1]) | Pimasertib 30 mg (All Regimens [Part 1]) | Pimasertib 42 mg (All Regimens [Part 1]) | Pimasertib 45 mg (All Regimens [Part 1]) | Pimasertib 60 mg (All Regimens [Part 1]) | Pimasertib 75 mg (All Regimens [Part 1]) | Pimasertib 90 mg (All Regimens [Part 1])
Number analyzed (Participants) | 11 | 10 | 8 | 9 | 13 | 2 | 16 | 5 | 1
nanogram/milliliter | 23.6 (40.1) | 59.3 (53.1) | 69.6 (39.2) | 150.1 (63.7) | 187.8 (25.3) | 123.2 (63.4) | 231.4 (48.2) | 383.2 (57.6) | 486.3 (NA) — Geometric coefficient of variation was not available as only 1 subject was evaluated for this group

6. Secondary Outcome: Part 1: Time to Reach Maximum Plasma Concentration (Tmax): Single Dose
Time Frame: Predose 0.5, 1.0, 1.5, 2.0, 2.5, 4.0, 6.0, and 10.0 hours post-dose on Day 1 of cycle 1; Regimen 1, 2 and 3
Population: Pharmacokinetic analysis set included all the subjects who received at least 1 dose of trial medication and provided pharmacokinetic samples per protocol. N (number of subject analyzed) signifies subjects evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Pimasertib 8 mg (All Regimens [Part 1]) | Pimasertib 15 mg (All Regimens [Part 1]) | Pimasertib 23 mg (All Regimens [Part 1]) | Pimasertib 30 mg (All Regimens [Part 1]) | Pimasertib 42 mg (All Regimens [Part 1]) | Pimasertib 45 mg (All Regimens [Part 1]) | Pimasertib 60 mg (All Regimens [Part 1]) | Pimasertib 75 mg (All Regimens [Part 1]) | Pimasertib 90 mg (All Regimens [Part 1])
Number analyzed (Participants) | 9 | 7 | 9 | 7 | 9 | 4 | 19 | 10 | 4
hour | 0.94 (41.18) | 2.25 (53.20) | 1.56 (151.73) | 1.09 (38.74) | 1.11 (78.05) | 1.12 (19.62) | 1.03 (40.27) | 2.70 (96.84) | 1.17 (76.62)

7. Secondary Outcome: Part 1: Time to Reach Maximum Plasma Concentration (Tmax): Multiple Dose
Time Frame: as for outcome 5
Population: Pharmacokinetic analysis set included all the subjects who received at least 1 dose of trial medication and provided pharmacokinetic samples per protocol. Number of subjects analysed refer to the subjects evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Pimasertib 8 mg (All Regimens [Part 1]) | Pimasertib 15 mg (All Regimens [Part 1]) | Pimasertib 23 mg (All Regimens [Part 1]) | Pimasertib 30 mg (All Regimens [Part 1]) | Pimasertib 42 mg (All Regimens [Part 1]) | Pimasertib 45 mg (All Regimens [Part 1]) | Pimasertib 60 mg (All Regimens [Part 1]) | Pimasertib 75 mg (All Regimens [Part 1]) | Pimasertib 90 mg (All Regimens [Part 1])
Number analyzed (Participants) | 11 | 10 | 8 | 9 | 13 | 2 | 16 | 5 | 1
hour | 1.44 (78.61) | 1.75 (83.12) | 2.03 (59.04) | 1.99 (70.40) | 1.64 (73.93) | 1.41 (52.11) | 1.78 (112.59) | 2.75 (21.83) | 2.00 (NA) — Geometric coefficient of variation was not available as only 1 subject was evaluated for this group.

8. Secondary Outcome: Part 1: Apparent Terminal Half-Life (t1/2) of Pimasertib: Single Dose
Description: The apparent terminal half-life was defined as the time required for the plasma concentration of drug to decrease 50% in the final stage of its elimination.
Time Frame: Predose 0.5, 1.0, 1.5, 2.0, 2.5, 4.0, 6.0, and 10.0 hours post-dose on Day 1 of cycle 1; Regimen 1, 2 and 3
Population: Pharmacokinetic analysis set included all the subjects who received at least 1 dose of trial medication and provided pharmacokinetic samples. N (number of subject analyzed) signifies subjects evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Pimasertib 8 mg (All Regimens [Part 1]) | Pimasertib 15 mg (All Regimens [Part 1]) | Pimasertib 23 mg (All Regimens [Part 1]) | Pimasertib 30 mg (All Regimens [Part 1]) | Pimasertib 42 mg (All Regimens [Part 1]) | Pimasertib 45 mg (All Regimens [Part 1]) | Pimasertib 60 mg (All Regimens [Part 1]) | Pimasertib 75 mg (All Regimens [Part 1]) | Pimasertib 90 mg (All Regimens [Part 1])
Number analyzed (Participants) | 9 | 4 | 6 | 7 | 8 | 4 | 18 | 5 | 3
hour | 5.28 (41.55) | 3.52 (19.75) | 3.05 (13.96) | 4.01 (36.61) | 3.88 (42.26) | 3.45 (23.80) | 2.97 (21.92) | 4.21 (92.04) | 3.39 (49.59)

9. Secondary Outcome: Part 1: Apparent Terminal Half-Life (t1/2) of Pimasertib: Multiple Dose
Description: as for outcome 8
Time Frame: as for outcome 5
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Pimasertib 8 mg (All Regimens [Part 1]) | Pimasertib 15 mg (All Regimens [Part 1]) | Pimasertib 23 mg (All Regimens [Part 1]) | Pimasertib 30 mg (All Regimens [Part 1]) | Pimasertib 42 mg (All Regimens [Part 1]) | Pimasertib 45 mg (All Regimens [Part 1]) | Pimasertib 60 mg (All Regimens [Part 1]) | Pimasertib 75 mg (All Regimens [Part 1]) | Pimasertib 90 mg (All Regimens [Part 1])
Number analyzed (Participants) | 9 | 7 | 6 | 6 | 11 | 2 | 11 | 2 | 1
hour | 6.97 (75.47) | 10.91 (590.54) | 3.69 (22.69) | 3.93 (32.17) | 3.71 (21.38) | 3.96 (17.24) | 4.52 (66.99) | 8.44 (175.10) | 5.04 (NA) — Geometric coefficient of variation was not available as only 1 subject was evaluated for this group

10. Secondary Outcome: Part 1: Area Under Curve From Time Zero to Last Sampling Time at Which the Concentration is at or Above Lower Limit of Quantification (AUC0-t) of Pimasertib: Single Dose
Time Frame: Predose 0.5, 1.0, 1.5, 2.0, 2.5, 4.0, 6.0, and 10.0 hours post-dose on Day 1 of cycle 1; Regimen 1, 2 and 3
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter
Arm/Group | Pimasertib 8 mg (All Regimens [Part 1]) | Pimasertib 15 mg (All Regimens [Part 1]) | Pimasertib 23 mg (All Regimens [Part 1]) | Pimasertib 30 mg (All Regimens [Part 1]) | Pimasertib 42 mg (All Regimens [Part 1]) | Pimasertib 45 mg (All Regimens [Part 1]) | Pimasertib 60 mg (All Regimens [Part 1]) | Pimasertib 75 mg (All Regimens [Part 1]) | Pimasertib 90 mg (All Regimens [Part 1])
Number analyzed (Participants) | 9 | 6 | 9 | 7 | 9 | 4 | 19 | 10 | 4
hour*nanogram/milliliter | 54.0 (57.2) | 125.4 (42.4) | 230.9 (60.9) | 456.2 (25.5) | 581.8 (45.4) | 735.2 (47.2) | 863.8 (52.8) | 905.0 (92.8) | 1268.2 (31.9)

11. Secondary Outcome: Part 1: Area Under Curve From Time Zero to Last Sampling Time at Which the Concentration is at or Above Lower Limit of Quantification (AUC0-t) of Pimasertib: Multiple Dose
Time Frame: as for outcome 5
Population: Pharmacokinetic analysis set included all the subjects who received at least 1 dose of trial medication and provided pharmacokinetic samples. '"n" =Subjects evaluable for this outcome measure for specified categories for each reporting group, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter
Arm/Group | Pimasertib 8 mg (All Regimens [Part 1]) | Pimasertib 15 mg (All Regimens [Part 1]) | Pimasertib 23 mg (All Regimens [Part 1]) | Pimasertib 30 mg (All Regimens [Part 1]) | Pimasertib 42 mg (All Regimens [Part 1]) | Pimasertib 45 mg (All Regimens [Part 1]) | Pimasertib 60 mg (All Regimens [Part 1]) | Pimasertib 75 mg (All Regimens [Part 1]) | Pimasertib 90 mg (All Regimens [Part 1])
Number analyzed (Participants) | 11 | 10 | 8 | 9 | 13 | 2 | 16 | 5 | 1
hour*nanogram/milliliter | 131.4 (45.5) | 307.2 (75.4) | 321.9 (29.9) | 679.4 (53.7) | 761.2 (35.5) | 628.0 (28.2) | 991.6 (66.1) | 2195.2 (97.3) | 2144.7 (NA) — Geometric coefficient of variation was not available as only 1 subject was evaluated for this group.

12. Secondary Outcome: Part 1: Area Under Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Pimasertib: Single Dose
Description: The AUC0-inf was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity. It is obtained from AUC0-t plus AUCt-infinity.
Time Frame: Predose 0.5, 1.0, 1.5, 2.0, 2.5, 4.0, 6.0, and 10.0 hours post-dose on Day 1 of cycle 1; Regimen 1, 2 and 3
Population: Pharmacokinetic analysis set included all the subjects who received at least 1 dose of trial medication and provided pharmacokinetic samples. 'N'(number of subjects analyzed)=subjects evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter
Arm/Group | Pimasertib 8 mg (All Regimens [Part 1]) | Pimasertib 15 mg (All Regimens [Part 1]) | Pimasertib 23 mg (All Regimens [Part 1]) | Pimasertib 30 mg (All Regimens [Part 1]) | Pimasertib 42 mg (All Regimens [Part 1]) | Pimasertib 45 mg (All Regimens [Part 1]) | Pimasertib 60 mg (All Regimens [Part 1]) | Pimasertib 75 mg (All Regimens [Part 1]) | Pimasertib 90 mg (All Regimens [Part 1])
Number analyzed (Participants) | 9 | 4 | 6 | 7 | 8 | 4 | 18 | 5 | 3
hour*nanogram/milliliter | 80.5 (52.9) | 145.2 (42.1) | 315.6 (76.3) | 562.1 (33.3) | 734.9 (49.7) | 858.4 (49.6) | 1027.4 (49.2) | 1530.7 (135.3) | 1873.9 (68.8)

13. Secondary Outcome: Part 1: Area Under Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Pimasertib: Multiple Dose
Description: as for outcome 12
Time Frame: as for outcome 5
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter
Arm/Group | Pimasertib 8 mg (All Regimens [Part 1]) | Pimasertib 15 mg (All Regimens [Part 1]) | Pimasertib 23 mg (All Regimens [Part 1]) | Pimasertib 30 mg (All Regimens [Part 1]) | Pimasertib 42 mg (All Regimens [Part 1]) | Pimasertib 45 mg (All Regimens [Part 1]) | Pimasertib 60 mg (All Regimens [Part 1]) | Pimasertib 75 mg (All Regimens [Part 1]) | Pimasertib 90 mg (All Regimens [Part 1])
Number analyzed (Participants) | 9 | 7 | 6 | 6 | 11 | 2 | 11 | 2 | 1
hour*nanogram/milliliter | 226.2 (91.0) | 789.3 (1038.0) | 451.2 (39.4) | 1030.2 (51.6) | 938.0 (46.6) | 786.7 (21.2) | 1270.8 (104.3) | 2712.6 (456.7) | 2830.7 (NA) — Geometric coefficient of variation was not available as only 1 subject was evaluated for this group.

14. Secondary Outcome: Part 1: Apparent Oral Clearance (CL/f) of Pimasertib: Single Dose
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Apparent clearance after oral dose (CL/f) is influenced by the fraction absorbed. Data for Pimasertib 75 mg arm was not available for all the regimens combined, thus reported as separate outcome measure and not included in this outcome.
Time Frame: Predose 0.5, 1.0, 1.5, 2.0, 2.5, 4.0, 6.0, and 10.0 hours post-dose on Day 1 of cycle 1; Regimen 1, 2 and 3
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour
Arm/Group | Pimasertib 8 mg (All Regimens [Part 1]) | Pimasertib 15 mg (All Regimens [Part 1]) | Pimasertib 23 mg (All Regimens [Part 1]) | Pimasertib 30 mg (All Regimens [Part 1]) | Pimasertib 42 mg (All Regimens [Part 1]) | Pimasertib 45 mg (All Regimens [Part 1]) | Pimasertib 60 mg (All Regimens [Part 1]) | Pimasertib 90 mg (All Regimens [Part 1])
Number analyzed (Participants) | 9 | 4 | 6 | 7 | 8 | 4 | 18 | 3
liter/hour | 99.43 (52.86) | 103.29 (42.07) | 72.88 (76.28) | 53.37 (33.26) | 57.15 (49.72) | 52.42 (49.59) | 58.40 (49.21) | 48.03 (68.78)

15. Secondary Outcome: Part 1: Apparent Oral Clearance (CL/f) of Pimasertib for Pimasertib 75 mg Reporting Arm: Single Dose
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Apparent clearance after oral dose (CL/f) is influenced by the fraction absorbed.
Time Frame: Predose 0.5, 1.0, 1.5, 2.0, 2.5, 4.0, 6.0, and 10.0 hours post-dose on Day 1 of cycle 1; Regimen 1, 2 and 3
Population: Pharmacokinetic analysis set included all the subjects who received at least 1 dose of trial medication and provided pharmacokinetic samples. 'N'(number of subjects analyzed)=subjects evaluable for this measure and "n" = subjects evaluable for the specified regimen.
Measure: Mean (Standard Deviation); unit: liter/hour
Arm/Group | Pimasertib 75 mg (All Regimens [Part 1])
Number analyzed (Participants) | 4
liter/hour
  Regimen 1 (n=0) | NA (NA) — For Regimen 1, number of subjects analyzed = 0 as no subject received 75 mg dose.
  Regimen 2 (n=3) | 93 (103.367)
  Regimen 3 (n=1) | 45 (NA) — Standard Deviation could not be estimated as there was only 1 participant assessed for the specified category.

16. Secondary Outcome: Part 1: Apparent Oral Clearance (CL/f) of Pimasertib: Multiple Dose
Description: as for outcome 15
Time Frame: as for outcome 5
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour
Arm/Group | Pimasertib 8 mg (All Regimens [Part 1]) | Pimasertib 15 mg (All Regimens [Part 1]) | Pimasertib 23 mg (All Regimens [Part 1]) | Pimasertib 30 mg (All Regimens [Part 1]) | Pimasertib 42 mg (All Regimens [Part 1]) | Pimasertib 45 mg (All Regimens [Part 1]) | Pimasertib 60 mg (All Regimens [Part 1]) | Pimasertib 75 mg (All Regimens [Part 1]) | Pimasertib 90 mg (All Regimens [Part 1])
Number analyzed (Participants) | 11 | 9 | 8 | 7 | 12 | 2 | 13 | 4 | 1
liter/hour | 60.90 (45.51) | 46.74 (78.85) | 66.52 (33.40) | 37.95 (47.59) | 55.80 (35.90) | 69.23 (33.40) | 65.11 (65.69) | 34.44 (119.51) | 41.96 (NA) — Geometric coefficient of variation was not available as only 1 subject was evaluated for this group.

17. Secondary Outcome: Part 1: Apparent Oral Volume of Distribution (Vz/f) of Pimasertib:Single Dose
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Apparent volume of distribution after oral dose (Vz/f) was influenced by the fraction absorbed. Data for Pimasertib 75 mg arm was not available for all the regimens combined, thus reported as separate outcome measure and not included in this outcome.
Time Frame: Predose 0.5, 1.0, 1.5, 2.0, 2.5, 4.0, 6.0, and 10.0 hours post-dose on Day 1 of cycle 1; Regimen 1, 2 and 3
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Pimasertib 8 mg (All Regimens [Part 1]) | Pimasertib 15 mg (All Regimens [Part 1]) | Pimasertib 23 mg (All Regimens [Part 1]) | Pimasertib 30 mg (All Regimens [Part 1]) | Pimasertib 42 mg (All Regimens [Part 1]) | Pimasertib 45 mg (All Regimens [Part 1]) | Pimasertib 60 mg (All Regimens [Part 1]) | Pimasertib 90 mg (All Regimens [Part 1])
Number analyzed (Participants) | 9 | 4 | 6 | 7 | 8 | 4 | 18 | 3
liter | 757.5 (48.3) | 524.8 (51.5) | 320.8 (60.1) | 308.8 (27.1) | 320.2 (40.4) | 260.8 (46.9) | 250.3 (48.5) | 235.2 (24.2)

18. Secondary Outcome: Part 1: Apparent Oral Volume of Distribution (Vz/f) of Pimasertib for Pimasertib 75 mg Reporting Arm:Single Dose
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Apparent volume of distribution after oral dose (Vz/f) was influenced by the fraction absorbed.
Time Frame: Predose 0.5, 1.0, 1.5, 2.0, 2.5, 4.0, 6.0, and 10.0 hours post-dose on Day 1 of cycle 1; Regimen 1, 2 and 3
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Pimasertib 75 mg (All Regimens [Part 1])
Number analyzed (Participants) | 4
liter
  Regimen 1 (n = 0) | NA (NA) — For Regimen 1, number of subjects analyzed = 0 as no subject received 75 mg dose.
  Regimen 2 (n = 3) | 442.2 (214.6)
  Regimen 3 (n = 1) | 196.0 (NA) — Standard Deviation could not be estimated as there was only 1 participant assessed for the specified category.

19. Secondary Outcome: Part 1: Apparent Oral Volume of Distribution (Vz/f) of Pimasertib: Multiple Dose
Description: as for outcome 18
Time Frame: as for outcome 5
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Pimasertib 8 mg (All Regimens [Part 1]) | Pimasertib 15 mg (All Regimens [Part 1]) | Pimasertib 23 mg (All Regimens [Part 1]) | Pimasertib 30 mg (All Regimens [Part 1]) | Pimasertib 42 mg (All Regimens [Part 1]) | Pimasertib 45 mg (All Regimens [Part 1]) | Pimasertib 60 mg (All Regimens [Part 1]) | Pimasertib 75 mg (All Regimens [Part 1]) | Pimasertib 90 mg (All Regimens [Part 1])
Number analyzed (Participants) | 9 | 7 | 6 | 6 | 11 | 2 | 11 | 2 | 1
liter | 601.7 (79.2) | 863.7 (193.5) | 332.8 (14.5) | 207.8 (46.8) | 293.1 (27.6) | 395.1 (52.9) | 422.0 (79.2) | 689.9 (16.0) | 305.2 (NA) — Geometric coefficient of variation was not available as only 1 subject was evaluated for this group.

20. Secondary Outcome: Part 1: Percentage of Subjects With Best Overall Response
Description: The best overall response was reported as either of the following: (1) Morphologic complete remission (CR) = normalization of the peripheral blood absolute neutrophil count (PBANC) >1.0x10^9 per liter (/L), platelets >100x10^9 /L, bone marrow aspirate with less than or equal to (<=) 5 percent (%) blasts, no blasts with Auer rods (AML only). (2) Complete remission with incomplete blood count recovery (CRi) = Same as CR without normalization of PBANC and platelet count. (3) Partial remission (PR) = normalization of PBANC >1.0x10^9/L, platelets >100x10^9/L, and at least a 50% decrease in the percentage of marrow aspirate blasts to 5-25%, or marrow blasts less than (<) 5%. (4) Progressive disease (PD) = >50% increase in peripheral blood or bone marrow blasts. (5) Stable disease (SD) = Subjects who failed to achieve CR, CRi or PR and without criteria for PD.
Time Frame: Day 29 of every alternate 29-day cycle until progression reported between day of first subject randomized, September 2009, until cut-off date, December 2012
Population: The efficacy analysis set included all subjects who received at least 1 administration of planned dose of pimasertib and had at least 1 efficacy assessment after the first dose. 'N' (number of subjects analyzed)=subjects evaluable for this outcome measure.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Regimen 1 (Part 1) | Regimen 2 (Part 1) | Regimen 3 (Part 1)
Number analyzed (Participants) | 20 | 22 | 7
Percentage of Subjects
  CR | 0.0 | 0.0 | 0.0
  CRi | 0.0 | 0.0 | 0.0
  PR | 0.0 | 0.0 | 0.0
  SD | 60.0 | 77.3 | 71.4
  PD | 40.0 | 22.7 | 28.6

21. Secondary Outcome: Part 2: Number of Subjects With TEAEs, Serious TEAEs, TEAEs Leading to Death and TEAEs Leading to Permanent Treatment Discontinuation
Description: An adverse event (AE) was defined as any new untoward medical occurrences/worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that results in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect.
Time Frame: Up to 3 years
Population: This outcome measure was not analyzed as the trial was terminated during safety run-in (Part 1).
Arm/Group | Regimen 1 (Part 2) | Regimen 2 (Part 2)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. SAEs and Other AEs (non-SAEs) were reported.
Arm/Group | Regimen 1 (Part 1) | Regimen 2 (Part 1) | Regimen 3 (Part 1)
Serious Adverse Events (participants affected / at risk) | 24/33 | 28/32 | 12/15
Other Adverse Events (participants affected / at risk) | 32/33 | 30/32 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen 1 (Part 1) (N=33) | Regimen 2 (Part 1) (N=32) | Regimen 3 (Part 1) (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 | 9 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Photopsia (Eye disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Caecitis (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Asthenia (General disorders) | 0 | 1 | 1
Disease progression (General disorders) | 0 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 5 | 1
Bacteraemia (Infections and infestations) | 2 | 2 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 3 | 0
Clostridial infection (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0
Human herpes virus 6 infection (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Lung Infection (Infections and infestations) | 2 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 7 | 4 | 3
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 3 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Asparatate aminotransferase increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0
White Blood Cell Count Increased (Investigations) | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1
Subdural hygroma (Nervous system disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Nephritic syndrome (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 1 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen 1 (Part 1) (N=33) | Regimen 2 (Part 1) (N=32) | Regimen 3 (Part 1) (N=15)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Pneumopericardium (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 1 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0
Chorioretinopathy (Eye disorders) | 0 | 3 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0
Conjunctival oedema (Eye disorders) | 0 | 1 | 1
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 1 | 0
Erythema of eyelid (Eye disorders) | 1 | 0 | 0
Eyelid disorder (Eye disorders) | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 1
Lacrimation increased (Eye disorders) | 0 | 1 | 0
Macular Degeneration (Eye disorders) | 0 | 1 | 1
Macular oedema (Eye disorders) | 1 | 0 | 0
Metamorphopsia (Eye disorders) | 0 | 1 | 0
Ocular hypertension (Eye disorders) | 1 | 0 | 0
Optic disc haemorrhage (Eye disorders) | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 1 | 2 | 0
Photopsia (Eye disorders) | 0 | 2 | 0
Retinal detachment (Eye disorders) | 2 | 4 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 2
Retinal oedema (Eye disorders) | 0 | 0 | 1
Retinal vein occlusion (Eye disorders) | 1 | 0 | 0
Scotoma (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 4 | 5 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 2 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0
Xerophthalmia (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 14 | 16 | 8
Dry mouth (Gastrointestinal disorders) | 2 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 2 | 1
Gingival inflammation (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 1 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 4 | 2 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 10 | 7 | 2
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1
Stomatitis necrotising (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 6 | 1
Asthenia (General disorders) | 4 | 5 | 2
Chest pain (General disorders) | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 0
Face oedema (General disorders) | 0 | 1 | 2
Fatigue (General disorders) | 5 | 5 | 2
Generalised oedema (General disorders) | 1 | 0 | 0
Hyperthermia (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 1
Malaise (General disorders) | 1 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 6 | 8 | 4
Pyrexia (General disorders) | 7 | 8 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Graft versus host disease in intestine (Immune system disorders) | 0 | 1 | 0
Graft versus host disease in skin (Immune system disorders) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 2 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Herpes simplex ophthalmic (Infections and infestations) | 1 | 0 | 0
Human herpesvirus 6 virus infection (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 2 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Eschar (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 2 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 3 | 0 | 1
Alanine aminotransferase increased (Investigations) | 6 | 4 | 1
Aspartate aminotransferase increased (Investigations) | 8 | 7 | 3
Blood albumin decreased (Investigations) | 4 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 5 | 3 | 2
Blood bilirubin increased (Investigations) | 2 | 0 | 0
Blood calcium decreased (Investigations) | 4 | 2 | 0
Blood creatine increased (Investigations) | 0 | 1 | 1
Blood creatinine (Investigations) | 1 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 1
Blood glucose increased (Investigations) | 2 | 1 | 1
Blood magnesium decreased (Investigations) | 2 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 1
Blood sodium decreased (Investigations) | 4 | 1 | 0
Blood urea increased (Investigations) | 0 | 1 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 3 | 0 | 1
Haemoglobin decreased (Investigations) | 2 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 3 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 5 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Aphonia (Nervous system disorders) | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 7 | 5 | 2
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 6 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Hypokinesia (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 2 | 0
Agitation (Psychiatric disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 1 | 1
Confusional state (Psychiatric disorders) | 3 | 3 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 2 | 1
Dysuria (Renal and urinary disorders) | 2 | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0 | 1
Testis discomfort (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 6 | 4
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 1
Hypotension (Vascular disorders) | 4 | 6 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
Infusion site oedema (General disorders) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The trial has been terminated due to an estimated low probability of clinical benefit based on limited anti-leukemic effects observed in safety run-in (Part 1).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other